CLINICAL TRIAL: NCT02870530
Title: Single Anastomosis Sleeve Jejunal (SAS-J) Bypass as A Treatment for Morbid Obesity
Brief Title: Single Anastomosis Sleeve Jejunal (SAS-J) Bypass
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Alaa Mstafa Hassan Sewefy, MD, Lecturer & consultant of general surgery, Department of surgery, Minia university hospital, Egypt, Minia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: fac.med.016
Record Dates: First submitted 2016-08-10; First posted 2016-08-17 (Estimated); Last update posted 2022-03-11 (Actual); Status verified 2022-02

CONDITIONS: Morbid Obesity
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Anastomosis Sleeve Jejunal (SAS-J) Bypass (Experimental): Single Anastomosis Sleeve Jejunal (SAS-J) Bypass as A treatment for Morbid
  Interventions: Procedure: Single Anastomosis Sleeve Jejunal (SAS-J) Bypass

INTERVENTIONS:
Procedure: Single Anastomosis Sleeve Jejunal (SAS-J) Bypass — Single Anastomosis Sleeve Jejunal (SAS-J) Bypass as A treatment for Morbid

SUMMARY:
The purpose of this study is to determine the efficacy of single anastomoses sleeve jejunal bypass as a treatment for morbid obesity

DETAILED DESCRIPTION:
in this study the investigators aim to test a new technique ( single anastomoses sleeve jejunal as a treatment for morbid obesity Which is a modification of Single anastomoses sleeve ileal bypass with short biliary limb ( about one third of the small intestine from the Duodeno-jejunal junction

ELIGIBILITY:
Inclusion Criteria:

* obese patients with BMI more than 40
* patients fit for laparoscopic surgery
* give approval to share in the study

Exclusion Criteria:

* patients refused to share in the study
* patients unfit for surgery
* patients aged less than 18 and older than 50
* patients with BMI less than 50
* patient with previous upper abdominal surgery either for obesity or other diseases
* patients with preoperative GERD clinically or by investigation

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2016-11; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
operative time | the 1st 24 hours
  the operative time from skin incision to skin closure
intraoperative complications | the 1st 24 hours
  intraoperative complications like bleeding, other organs injuries
the postoperative weight loss | 12 month
  the percentage of weight loss from total excess body weight

SECONDARY OUTCOMES:
effect on metabolic syndrome if present | 12 months
  effect on blood sugar level, blood pressure and blood cholesterol level

OTHER OUTCOMES:
postoperative biliary reflux | 3 months
  the presence of postoperative biliary reflux clinically and by upper endoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Alaa M Sewefy, MD, Study Chair — Lecturer & consultant of general surgery, Department of surgery, Minia university hospital, Egypt.
Locations (1):
- Minia university hospital, Minya, Egypt

IPD SHARING:
Plan to Share IPD: Undecided